CLINICAL TRIAL: NCT00278083
Title: A Randomised, Double Blind, Placebo-controlled, Parallel Group Pilot Study to Determine the Effect of REMICADE on Safety, Efficacy and Biomarkers of Inflammation in Patients With Asthma Receiving Inhaled Corticosteroids
Brief Title: TNF-alpha Directed Therapy in Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C0168T42
Record Dates: First submitted 2006-01-17; First posted 2006-01-18 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Asthma
Keywords: Pharmacology; Asthma; TNF-alpha
MeSH Terms: conditions — Asthma | interventions — Respiratory Physiological Phenomena; Blood Specimen Collection; Urinalysis

INTERVENTIONS:
Drug: Study drug administration
Procedure: Tuberculin intradermal skin test
Procedure: Lung function test for FEV1
Procedure: Asthma symptom scores diary
Procedure: Quality of life diary
Procedure: Breath nitric oxide
Procedure: Breath condensate
Procedure: Sputum induction
Procedure: Blood sampling
Procedure: Urinalysis

SUMMARY:
This trial is a randomised, single-center, placebo-controlled, double blind, parallel group study in patients with asthma symptomatic on inhaled steroids.

This trial will examine the efficacy and safety of 5 mg/kg doses of infliximab in patients with inhaled corticosteroid-dependent asthma. The primary objective of this study is to obtain pharmacological evidence for a role of the pro-inflammatory cytokine TNF-alpha in patients with asthma symptomatic on inhaled steroids and to evaluate the safety and tolerability of repeated intravenous administration of infliximab.

DETAILED DESCRIPTION:
Study Overview This trial is a randomised, single-center, placebo-controlled, double blind, parallel group study in patients with asthma symptomatic on inhaled steroids.

Patient Population Patients eligible for this study will have a diagnosis of moderate asthma defined by the American Thoracic Society criteria for > 1 year. These patients should be taking inhaled steroids at doses equivalent to </= 400µg and </= 2000µg per day beclomethasone diproprionate but not oral steroid medication. Patients taking additional oral steroids are required to stop oral medication at least one month prior to pre-screening.

Many of these patients will be receiving long-acting beta2-agonists and this therapy will be discontinued for 48h before starting the run-in. In addition, the following therapies are not allowed: 1) anticholinergics; 2) theophylline; 3) oral beta2-agonists; 4) antihistamines; 5) inhaled cromolyn sodium or nedocromil; 6) leukotriene antagonists.

Patients using these prohibited medications will be asked to discontinue use 2 weeks prior to the screening examination. During this washout period, patients will keep a clinical diary and will remain in contact with the clinical research center.

Eligible patients for screening will maintain stable doses of their normal inhaled steroids in doses equivalent to >/= 400 µg and </= 2000µg per day beclomethasone diproprionate and will be able to use short-acting beta2-agonists for symptom relief.

Screening At screening, eligible patients will have a baseline screening FEV1 of >/= 60 to </= 90% of predicted at least 4 hours after the last usage of a short-acting beta2-agonist. Patients will have reversible airway obstruction: a >/= 12% increase in FEV1 in comparison to baseline should be shown within 30 minutes after taking 200 µg salbutamol. If airway reversibility cannot be demonstrated during this visit, patients are eligible for re-testing. Reversible airway disease may be demonstrated at any time between screening and start of run-in period. The 2 to 4 week run-in period will start immediately after demonstration of reversible lung disease.

Patients will also have skin tests to a standard battery of bronchial allergens performed at screening. Patients should have both a purified protein derivative (PPD) skin test and a chest radiograph prior to their first infusion. Patients with evidence of either latent or active tuberculosis (TB) will not be enrolled.

Run-in Period Following acceptable screening tests patients will complete a baseline run-in of 2 to 4 weeks duration prior to the study start. During this period patients will be required to keep a symptom diary and to record baseline lung function parameters using an electronic spirometer. As before, patients will be maintained on their normal inhaled steroids in doses equivalent to >/= 400 µg and </= 2000µg per day beclomethasone diproprionate and will be able to use short-acting beta2-agonists for symptom relief. No other asthma medications will be allowed during this period and the rest of the study. Use of all other, non-asthma, medication will be reviewed by the Investigator and allowed at his/her discretion provided a stable dose regimen is maintained where possible throughout the study.

Baseline Visit (day -1) The day before the first drug administration, patients will attend the clinical research unit and diary cards will be reviewed. In order to enter the study the patients must have a mean total daily symptom score >/= 4 measured during the last 7 days of the baseline run-in period [A symptom scale with scores ranging from 0 (=symptom free) to 3 (=severe symptoms) is used, with 6 questions, and a total maximum daily symptom score of 18, see appendix D)] and/or have a >/= 10% and < 30% diurnal variation in PEFR measured on at least 2 of 7 days during the same period.

Diurnal variation in PEFR is defined from morning and evening PEFR values; in the morning and evening the PEFR is determined on 3 immediately consecutive occasions and the highest value taken. The calculation of diurnal variation is based on:

[(higher (am or pm) PEFR- lower (am or pm) PEFR) / higher (am or pm) PEFR x 100].

In eligible patients, the following pharmacodynamic assessments will be made: breath NO levels (non-nasal) and breath condensates, pulmonary function testing (FEV1, FVC and PEFR), sputum induction for markers of inflammation, and a blood sample collection for the measurement of markers of inflammation.

Study Treatments Patients will be randomised in a 1:1 ratio to treatment with infliximab or placebo, respectively. PRI will provide the randomisation list. At t=0 weeks, patients will either receive 5 mg/kg infliximab (Group I, n=20) or placebo (Group II, n=20). Subsequently, infliximab or placebo will be infused at weeks 2 and 6. Throughout the study period up to week 12, patients will be allowed to use inhaled corticosteroids at a stable dose regimen. Salbutamol, a short-acting beta2-agonist, will be allowed as necessary to relieve symptoms.

During the study, the two treatment groups are defined as:

Group I: Infliximab 5 mg/kg + short-acting beta2-agonist (as needed) + inhaled corticosteroids (equivalent to >/= 400 µg and </= 2000µg per day beclomethasone diproprionate).

Group II: Placebo + short-acting beta2-agonist (as needed) + inhaled corticosteroids (equivalent to >/= 400 µg and </= 2000µg per day beclomethasone diproprionate).

Study Evaluations Throughout the study, starting with the baseline run-in period, patients will be required to daily record their PEFR and FEV1 (morning and evening), short-acting beta2-agonist use and clinical symptoms using a diary card. Mean weekly scores will be calculated for each parameter starting at week -1 up to week 12. Prior to administration of study drug at week 0 and, in addition, at weeks 1, 8 and 12, the following pharmacodynamic assessments will be made: breath NO levels, breath condensate leukotriene B4 & C4, pulmonary function testing (FEV1, FVC and PEFR), sputum induction for markers of inflammation (weeks 0, 1 and 8 only) and levels of markers of inflammation in peripheral blood. In addition, at weeks 2 and 6, breath NO levels will be measured and pulmonary function testing will be performed.

Safety Safety evaluations will include measurement of vital signs during and immediately after (for 2 hours) the infusion of study medications and assessment of adverse events (AEs) at each of the evaluation visits. Additional vital signs and lung function measurements will be performed immediately after each infusion and at t = 1 and 2 hours post dose. Routine laboratory tests will be performed at screening, at day -1 and at weeks 2, 6, 8 and 12. During the study, the medical monitor will regularly review safety data.

Follow-up During the last visit in week 12 to the clinical research center, a follow-up examination, including a physical examination and blood and urine chemistry will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of moderate asthma as defined by the American Thoracic Society criteria (NIH, 1997) for > 1 year.
2. Men and women, >/= 18 to </= 60 years of age and within 60-140% of desirable height and weight range established by the 1983 Metropolitan Life Insurance Company standards.
3. Non-smoker for at least 1 year and less than a 10 pack year history of smoking.
4. Screening values for haematology, biochemistry and urinalysis should be within clinically acceptable limits for this patient group.
5. Chest radiograph at screening must show no evidence of malignancy, infection, or fibrosis. The chest radiographs should also show no apical scarring, cavitary lesions, or calcified granulomas, as evidence of past tuberculosis infections.
6. Serological assays for hepatitis B and C must be negative for active infection.

Exclusion Criteria:

1. Are pregnant, nursing, or planning a pregnancy within 12 months of enrolment.
2. Diagnosis of chronic obstructive pulmonary disease, cystic fibrosis or other significant respiratory disorder (excluding asthma).
3. Exacerbation of asthma symptoms requiring hospitalisation within the previous 12 weeks.
4. History of clinically significant seasonal allergies will require that the patient is studied outside the allergy season.
5. Have been previously treated with infliximab or any other therapeutic agent targeted at reducing TNF.
6. Have been treated with any anti-CD-4 antibody.
7. Have been treated with any investigational drug within the previous 3 months or within 5 half-lives, whichever is greater.
8. Have previously used cyclophosphamide, nitrogen mustard, chlorambucil, or other alkylating agents.
9. Have a history of any clinically significant adverse reaction to murine or chimeric proteins, including but not limited to allergic reactions.

11. Have had a serious infection during the previous 2 months. 12. Have a chronic or recurrent infectious disease 13. Have a history of opportunistic infections 14. Have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.

15. Have a history of lymphoproliferative disease, including lymphoma 16. Currently have any known malignancy or have a history of malignancy within the previous 5 years.

17. Have had substance abuse (drug or alcohol) problem within the previous 10 years.

18. Use of restricted respiratory medication prior to screening within the following time periods: 1) oral or systemic steroids, 1 month; 2) immunosuppressant therapy, 3 months.

19. Have a history of chronic cough, haemoptysis, weight loss, or pyrexia considered suggestive of possible current tuberculosis infection.

20. Patients with current active tuberculosis (TB) or atypical mycobacterial infection or a previous history of these infections.

21. Be considered at high risk for tuberculosis according to US Centers for Disease Control and Prevention (CDC) criteria, 22. A tuberculin (purified protein derivative, PPD) intradermal skin test > 10mm induration.

23. Have demyelinating disease (multiple sclerosis), autoimmune conditions such as systemic lupus.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 2001-10; Study Completion 2004-04

PRIMARY OUTCOMES:
Change from baseline (prior to visit 4: days -7 to -1) to week 8 (prior to visit 8: days 49-56) in mean morning PEFR from clinical diaries:
The morning PEFR for a 7 day period (week 7 to 8) will be compared to the 7 day period prior to first administration (days -7 to -1).

SECONDARY OUTCOMES:
1. Evening PEFR
2. FEV1 from clinical diaries and on study visits
3. Diurnal variation in PEFR
4. Symptoms score
5. Short-acting beta2-agonist usage = rescue salbutamol
6. Exacerbation's and episode-free days
7. Quality of life (St. George's Respiratory Questionnaire)
8. Exhaled breath NO and breath condensates
9. Sputum levels of IL-8, TNF-alpha and eotaxin (in supernatant) and differential white cell count
10. Peripheral blood eosinophil count, and total IgE
11. Expression of mRNA related to inflammation in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Trevor T Hansel, FRCPath PhD, Principal Investigator — Imperial College London
Locations (1):
- NHLI Clinical Studies Unit, London, United Kingdom